CLINICAL TRIAL: NCT06749496
Title: Evaluation of Delefilcon A and Senofilcon A Daily Disposable Toric Soft Contact Lenses Over One Week of Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6594
Record Dates: First submitted 2024-12-23; First posted 2024-12-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects will be randomized into the Test/Control sequence, to wear each study lens (Test lens and Control lens) in a daily disposable modality for approximately one week with a washout period of one week between study lens wear periods.
  Interventions: Device: Test Lens; Device: Control Lens
- Control/Test (Experimental): Eligible subjects will be randomized into the Control/Test sequence, to wear each study lens (Control lens and Test lens) in a daily disposable modality for approximately one week with a washout period of one week between study lens wear periods.
  Interventions: Device: Test Lens; Device: Control Lens

INTERVENTIONS:
Device: Test Lens — ACUVUE® OASYS MAX 1-Day for ASTIGMATISM (AOM1DfA).
Device: Control Lens — Alcon DAILIES TOTAL1® for Astigmatism Contact Lenses (DT1fA).

SUMMARY:
This is a prospective, multi-site, 4-visit, bilateral, dispensing, randomized, controlled, double-masked, 2x2 crossover study to evaluate subjective comfort, overall opinion and end of day comfort following wear of two different contact lenses.

ELIGIBILITY:
Potential subjects must satisfy all of the following criteria to be enrolled in the study:

The subject must:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e., not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 2 days per week during the past four weeks.
5. Possess a wearable pair of spectacles that provide correction for distance vision.
6. In both eyes, have refractive error suitable for correction with the range of toric contact lens powers available in this study:

   6.1 Sphere powers (DS) -1.50 through -4.00 (inclusive) in 0.25 steps 6.2 Cylinder powers (DC) -0.75 and -1.25 6.3 Axes (°) 170, 180, 10, 80, 90 and 100
7. Have best corrected monocular distance visual acuity of 20/25 or better in each eye.

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The subject must not:

1. Be currently pregnant or lactating.
2. Be diabetic.
3. Be currently using any ocular medications or have any ocular infection of any type.
4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g., rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g., SynergEyes, SoftPerm) within the past 6 months.
6. Be currently wearing monovision or multifocal contact lenses.
7. Be currently wearing lenses in an extended wear modality.
8. Have a history of strabismus or amblyopia.
9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.
11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcome: Comfort | Up to 1-week follow-up
  Comfort, with respect to contact lens wear, will be assessed using the individual questionnaire item: 'I could wear these contact lenses comfortably for as long as I wanted to'. This item will utilize an agreement scale of, 1: Strongly Disagree, 2: Disagree, 3: Neither Agree nor Disagree, 4: Agree and 5: Strongly Agree.

SECONDARY OUTCOMES:
Overall Opinion | Up to 1-week follow-up
  Overall opinion, with respect to the study contact lenses, will be evaluated using the individual questionnaire item 'Considering your experience with the study contact lenses, which statement best describes your overall opinion of these contact lenses?'. This item will utilize an excellence scale of, 1: Poor, 2: Fair, 3: Good, 4: Very Good and 5: Excellent.
Comfort at the End of the Day | Up to 1-week follow-up
  Comfort at the end of the day, with respect to contact lens wear, will be assessed using the individual questionnaire 'These lenses were very comfortable at the end of the day'. This item will utilize an agreement scale of, 1: Strongly Disagree, 2: Disagree, 3: Neither Agree nor Disagree, 4: Agree and 5: Strongly Agree.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (12):
- United States (12):
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Omega Vision Center, Longwood, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Kannarr Eye Care - 101 North Broadway, Pittsburg, Kansas
  - Birmingham Vision Care, Bloomfield Hills, Michigan
  - Complete Eye Care of Medina, Medina, Minnesota
  - Sacco Eye Group, Vestal, New York
  - Procare Vision Centers, Granville, Ohio
  - Professional Vision Care Inc. - Westerville, Westerville, Ohio
  - Optometry Group, PLLC, Memphis, Tennessee
  - Tyler Eye Associates, Tyler, Texas
  - Botetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu